CLINICAL TRIAL: NCT05626829
Title: Application of Tranilast as a Radiosensitizer in the Treatment of Radiotherapy Resistant Nasopharyngeal Carcinoma: a Phase II Clinical Study
Brief Title: Tranilast as a Radiosensitizer in Reradiation of Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jian Guan (Other)
Responsible Party: Sponsor-Investigator, Jian Guan, chief physician, Nanfang Hospital, Southern Medical University
Organization: Nanfang Hospital, Southern Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2022-270
Record Dates: First submitted 2022-07-31; First posted 2022-11-25 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Nasopharyngeal Carcinoma; Recurrent Cancer
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Recurrence | interventions — tranilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tranilast (Experimental): concurrent Tranilast 100mg 3 times per day
  Interventions: Drug: Tranilast

INTERVENTIONS:
Drug: Tranilast — Tranilast capsules 100mg 3 times per day when reradiation

SUMMARY:
Nasopharyngeal carcinoma is one of the high incidence head and neck cancer in Southeast Asia. Radiotherapy is the main treatment for nasopharyngeal carcinoma, and its response rate can reach 80~90%. However, for radiotherapy resistant patients with metastasis and recurrence, the survival prognosis decreased significantly, and the 5-year overall survival rate was only 20% - 40%. Tranilast is an anti-allergic drug, which is clinically used to treat bronchial asthma and can inhibit fibroblasts α- SMA and type I collagen expression. Through experiments in vivo and in vitro, the investigators' research group has proved that Tranilast can inhibit the activity of tumor related fibroblasts, reduce the radiotherapy resistance of nasopharyngeal carcinoma, and has the radiosensitizing effect of nasopharyngeal carcinoma. This result has been published in J exp Clin cancer res (if=11.16). The investigators plan to carry out the clinical transformation of basic research, carry out a prospective intervention phase II clinical trial, compare the objective remission rate of patients with recurrent nasopharyngeal carcinoma treated with previous radiotherapy, and explore the safety and effectiveness of using Tranilast as a radiotherapy sensitizer for radiotherapy to resist the treatment of nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Sign informed consent
2. At least 18 years old on the date of signing the informed consent
3. Previously received standard radical radiotherapy and chemotherapy
4. Recurrent nasopharyngeal carcinoma in situ or cervical lymph nodes confirmed by pathological biopsy and imaging examination
5. After multidisciplinary consultation, there was a clear indication for surgery, and the patient was informed and refused to accept surgical treatment 6）ECOG PS：0/1

7) Laboratory examination confirmed good organ function, which should be carried out within 10 days before the first treatment.

Exclusion Criteria:

1. After evaluation, it does not meet the indications of re-radiotherapy
2. unable to take oral medication
3. Pregnancy or lactation
4. Known allergy to Tranilast
5. Patients who are judged by the researcher as unsuitable to participate in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2024-07-20 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
the Effectiveness of Tranilast in reradiation of recurrent nasopharyngeal carcinoma | 12 weeks after Tranilast treatment
  we use the objective response rate (ORR), according to the RESIST v1.0

SECONDARY OUTCOMES:
the Safety of Tranilast in reradiation of recurrent nasopharyngeal | 12 weeks after Tranilast treatment
  treatment-related adverse events will be assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Guan Jian, Ph.D., Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Southern medical university, Guangzhou, Guangdong, China

DOCUMENTS (1):
  • Study Protocol (2022-11-01): https://cdn.clinicaltrials.gov/large-docs/29/NCT05626829/Prot_000.pdf